CLINICAL TRIAL: NCT04115449
Title: Effect of Intravenous Dexmedetomidine on Patient Discomfort in Laparoscopic Cholecystectomy Under Spinal Anesthesia. A Randomized Control Study.
Brief Title: Effect of Intravenous Dexmedetomidine on Patient Discomfort in Laparoscopic Cholecystectomy Under Spinal Anesthesia.
Acronym: RCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, Anesthesia and Intensive care clinical researcher, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBRI
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Pain
Keywords: dexmedetomidine, shoulder pain, spinal anesthesia.
MeSH Terms: conditions — Shoulder Pain | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized double blinded control study which will be conducted in department of anesthesia and surgical Intensive care unit at Theodor Bilharz Research Institute after approval by research ethics committee and patient informed consent. 40 patients will be enrolled in the study and divided into two groups either (Dexa group (D) or Control group (C).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded randomized control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexa group (Experimental): Spinal anaesthesia will be performed through the L3-4 interspace in the sitting position. After dural puncture with a 25 G Quincke needle, 3.5 ml of hyperbaric bupivacaine 0.5% solution with fentanyl 20 μg will be injected intrathecally. Than manintance dose of dexmedetomidine will be titrated from (0.2- 0.6 mcg /kg/ min) according to the patient discomfort.
  After turning the patient supine, level of sensory block will be assessed by the pinprick test using a 24-gauge hypodermic needle, while the motor block level will be assessed by the modified Bromage scale. Insufflation of gas will be done at the rate of 1.5 liters/min and the maximum abdominal pressure will be kept at 12 mmHg. Supplementary oxygen at 4 liters/min will be given with face mask.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Normal Saline as a placebo will be infused over a period of ten minutes then spinal anaesthesia will be performed through the L3-4 interspace in the sitting position. After dural puncture with a 25 G Quincke needle, 3.5 ml of hyperbaric bupivacaine 0.5% solution with fentanyl 20 μg will be injected intrathecally. Then the placebo will be titrated according to patient discomfort.
  After turning the patient supine, level of sensory block will be assessed by the pinprick test using a 24-gauge hypodermic needle, while the motor block level will be assessed by the modified Bromage scale.Insufflation of gas will be done at the rate of 1.5 liters/min and the maximum abdominal pressure will be kept at 12 mmHg. Supplementary oxygen at 4 liters/min will be given with face mask.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Injection dexmedetomidine 1 mcg /kg will be infused over a period of ten minutes
  Arms: Dexa group
Drug: normal saline — Normal Saline as a placebo will be infused over a period of ten minutes
  Arms: Control group

SUMMARY:
Laparoscopic cholecystectomy (LC) has been routinely performed under general anesthesia despite the several disadvantages of general anesthesia compared to regional anesthesia.

There are multiple reports that have been published regarding the feasibility of spinal anesthesia for LC associated with many problems such as referred shoulder pain secondary to intra-abdominal pneumoperitoneum; patient anxiety, pain, and discomfort; and inadequate sedation.The aim of our study is to prospectively observe the feasibility of using intravenous dexmedetomidine to abolish patient discomfort and shoulder pain, thus making the patient more comfortable without causing excessive sedation and respiratory depression.

DETAILED DESCRIPTION:
This is a prospective, randomized double blinded control study which will be conducted in department of anesthesia and surgical Intensive care unit at Theodor Bilharz Research Institute after approval by research ethics committee and patient informed consent. 40 patients will be enrolled in the study and divided into two groups 20 patients each ; either (Dexa group (D) or Control group (C).

Anesthesia Technique:

A preoperative assessment, including a history, physical examination, review of laboratory data, and assignment of ASA classification will be performed on all patients prior to the procedure. Anesthesia and procedural consent will be obtained.

After premedication with i.v. midazolam 2 mg , patients will be transferred to the operating theatre. Ringer's solution 500 ml will be given over 15 min, and patients will be premedicated with intravenous ondensetron 4 mg and intravenous atropine 0.2 mg.

IN DEXA GROUP:

Injection dexmedetomidine 1 mcg /kg will be infused over a period of ten minutes then Spinal anaesthesia will be performed through the L3-4 interspace in the sitting position. After dural puncture with a 25 G Quincke needle, 3.5 ml of hyperbaric bupivacaine 0.5% solution with fentanyl 20 μg will be injected intrathecally. Than manintance dose of dexmedetomidine will be titrated from (0.2- 0.6 mcg /kg/ min) according to the patient discomfort.In CONTROL GROUP:

Normal Saline as a placebo will be infused over a period of ten minutes then spinal anaesthesia will be performed through the L3-4 interspace in the sitting position. After dural puncture with a 25 G Quincke needle, 3.5 ml of hyperbaric bupivacaine 0.5% solution with fentanyl 20 μg will be injected intrathecally. Then the placebo will be titrated according to patient discomfort.

In BOTH GROUPS:

After turning the patient supine, level of sensory block will be assessed by the pinprick test using a 24-gauge hypodermic needle, while the motor block level will be assessed by the modified Bromage scale (0 = no paralysis; 1 = unable to raise extended leg; 2 = unable to flex knee; 3 = unable to flex ankle) and recorded 10 min after placement in the supine position. Insufflation of gas will be done at the rate of 1.5 liters/min and the maximum abdominal pressure will be kept at 12 mmHg. Supplementary oxygen at 4 liters/min will be given with face mask.Heart rate (HR), non-invasive mean blood pressure (MBP), and respiratory rate will be monitored preoperatively, during dexmedetomidine infusion, after completion of infusion i.e. before spinal anaesthesia, after spinal anaesthesia, during creation of pneumoperitoneum, thereafter every 10 minutes, after desufflation and on admission to Post Anaesthesia Care Unit (PACU) If the systolic arterial pressure decreased to below 90 mm Hg or if mean arterial pressure decreased (MAP) 20% from baseline, ephedrine bolous will be given i.v. If heart rate decreased to, 45 beats min, i.v. atropine 0.5 mg will be administered.

Discomfort and shoulder pain will be assessed either by verbal complaint by the patient or by facial and body expression. Supplemental doses of fentanyl 25 μg were given if the patient is discomfort or in pain.

Any patient shall be converted to general anesthesia at any time intraoperatively due to persistent pain or discomfort despite administration of intravenous analgesics or sedatives or surgical procedure related indication.

Data Collection

1. Age
2. Sex
3. BMI
4. ASA
5. Abdominal discomfort
6. Referred shoulder pain
7. Arterial Blood pressue
8. Heart rate
9. Intraoperative Nausea/vomiting
10. Respiratory depression is defined as respiratory rate < 8 bpm.
11. Supplement of fentanyl
12. Conversion to general anesthesia
13. The severity of pain will be graded as nil, mild, moderate and severe.
14. Sedation level will be evaluated according to a four-point rating scale. 1, Patient fully awake; 2, patient somnolent but responds to verbal commands; 3, patient somnolent but responds to tactile stimuli; 4, patient asleep but responds to pain
15. The overall degree of patient satisfaction will be assessed using a three-point scale (good, moderate, and bad) on the first postoperative day.
16. Time of complete regression of spinal anaesthesia,
17. Post-operative complications: Nausea and Vomiting (PONV), Urine retention and Postdural puncture headache.

Statistical analysis Statistical analysis will be per-formed using the GraphPadInStat software package (GraphPad, San Diego, CA).The categorical factors are represented by the number and frequency (%) of cases. The continuous variables will represented by measures of central frequency and standard error. The statistical analysis was done by using unpaired t-test and Chi-square. p< 0.05 was considered statistically significant.

This is fourty patients will be prospectively enrolled for each study of patients who had been diagnosed to be able to reject the null hypothesis that the population means of the groups are equal with Power calculations suggested that a minimum of 16 subjects per group was required to detect 10% difference in arterial pressure between groups (taking type I or α error of 5%, type II or β error of 20% and Standard Deviation=10). To be on a safer side, 20 patients were included in each group (n=20).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2.
* Patients undergoing elective laparoscopic Cholecystectomy with estimated pneumoperitoneum time of 60 to 90 min.

Exclusion Criteria:

* Pregnancy.
* Lactating women.
* Any contraindication to spinal anesthesia e.g. Bleeding diathesis, infection at the puncture site, patient on anticoagulants or preexisting neurological deficits in lower extremities.
* Patients on α2-adrenergic receptors antagonists, calcium channel blockers, or angiotensin-converting enzyme inhibitors.
* Patients known allergic to bupivacaine or dexmedetomidine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Intraopertive shoulder pain | 60-90 minutes
  The severity of pain will be graded as nil, mild, moderate and severe.

SECONDARY OUTCOMES:
Number of intraoperative hypoxic episodes | 60-90 minutes.
  (Spo2 ≤95 %)

OTHER OUTCOMES:
Number of intraopertive hypotensive episodes. | 60-90 minutes.
  mean blood pressure decreased by more than 20% of the baseline.
Length of stay in PACU | average 1 hour.
  monitoring of length of stay in PACU to determine whether it is prolonged or not.

CONTACTS AND LOCATIONS:
Overall Officials: Moshira S Mohamed, MD, Principal Investigator — Theodor Bilharz Research Institute; Hend F Hassan, MD, Study Chair — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data available for the participant will be: Age, Sex, BMI and ASA classification. these data will available for other researchers.
  other personal data won't be shared to ensure patient privacy.
Supporting Information: Study Protocol, SAP
Time Frame: 6 month to 1 year

REFERENCES:
- [Background] Donmez T, Erdem VM, Uzman S, Yildirim D, Avaroglu H, Ferahman S, Sunamak O. Laparoscopic cholecystectomy under spinal-epidural anesthesia vs. general anaesthesia: a prospective randomised study. Ann Surg Treat Res. 2017 Mar;92(3):136-142. doi: 10.4174/astr.2017.92.3.136. Epub 2017 Feb 24. PMID 28289667